CLINICAL TRIAL: NCT03750877
Title: Evaluation of Median and Paramedian Approach in Spinal Anesthesia in Elderly Patients
Brief Title: Median and Paramedian Approach in Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trabzon Kanuni Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyfi KARTAL, MD, Assistant professor, Trabzon Kanuni Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: +90
Record Dates: First submitted 2018-11-17; First posted 2018-11-23 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Geriatric Patients; Efficacy, Self
Keywords: median approach; paramedian approach; geriatric patient; spinal anesthesia

STUDY DESIGN:
Intervention Model Description: The aim of this study was to evaluate the success rate of median and paramedian approach in spinal anesthesia in geriatric patients, number of trials, number of attempts at another interval due to failure, duration of procedure, patient comfort, change to other method in case of failure and success rate. In the study, two groups were formed: the median approach and the paramedian approach.
Who Masked: Participant
Masking Description: the number of files from the volunteer participants were grouped into one group and the ones with double file numbers were included in the other group.
  participants do not know which group of patients to be in. Only practitioners know about the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- median approach (Active Comparator): Spinal anesthesia will be performed with a conventional median approach
  Interventions: Procedure: median approach; Procedure: paramedian approach
- paramedian approach (Active Comparator): Spinal anesthesia will be applied with a paramedian approach.
  Interventions: Procedure: median approach; Procedure: paramedian approach

INTERVENTIONS:
Procedure: median approach — spinal anesthesia with median approach; is the known classical method and it is aimed to reach the spinal area from the middle line.
  Other Names: classical approach
Procedure: paramedian approach — In spinal anesthesia with a paramedian approach, 1 cm lateral and 1 cm caudal to reach the spinal area.

SUMMARY:
Spinal anesthesia (SA) is frequently used as anesthesia in many surgeries such as lower abdominal, inguinal, urogenital, rectal and lower extremities.

Conventional median approach (MA) is preferred more frequently, although MA or paramedian approach (PA) is used in SA. Especially in geriatric patients due to degenerative changes Although we are told that degenerative changes are less affected in PA during SA in the geriatric age group, few studies have been conducted on the subject and we aimed to evaluate the superiority of the two methods.

DETAILED DESCRIPTION:
In our study, 100 cases were planned to be evaluated prospectively. Patients scheduled for surgery under spinal anesthesia will undergo routine spinal preparation. After routine motorization, patients will be treated with MA or PA.

MA will be performed in a conventional manner and PA will be performed by adding 1 cm lateral and 1 cm caudal from the planned vertebral space to 10-15 degree medial and cephal.

If one of the patients with MA or PA fails, despite three attempts, the other method will be tried by another specialist. If the procedure fails or there are not enough blocks, a different anesthesia method will be applied.

The data of the patients included in the study were evaluated by a different researcher other than the SA physician; demographic data of the cases, type of operation, MA or PA in SA and the number of repeated attempts / trials for the procedure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 70 years
* elective surgery under spinal anesthesia
* those who agreed to participate in the study
* Those with American Society of Anesthesiologists (ASA) 1-3

Exclusion Criteria:

* who use opioid or other non-steroidal anti-inflammatory drugs regularly
* who are allergic to a drug used in the study
* had contraindications for spinal anesthesia,
* drug addiction
* obese patients (Body Mass Index ≥ 35)
* migraine and chronic headache
* Spinal anesthesia can not be performed in more than 3 trials, but passed to the general anesthesia
* those who do not agree to participate in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-02-22 (Actual)

PRIMARY OUTCOMES:
spinal needle touches the spinal bone | during the procedure of spinal anesthesia
  The ability of getting a successful spinal anesthesia with a single skin puncture and no needle redirection.
Number of repeated attempts (attempts): | during the procedure of spinal anesthesia
  The ability of getting a successful spinal anesthesia with a single skin puncture and no needle redirection.
duration of procedure | during the procedure of spinal anesthesia
  In spinal anesthesia, the time to reach the skin and the spinal area will be evaluated.

SECONDARY OUTCOMES:
success rate of spinal needle insertion | during the procedure of spinal anesthesia
  The ability of getting a successful spinal anesthesia with a single skin puncture regardless of needle redirection.
Complications of the procedure | during the procedure of spinal anesthesia and 1 week after spinal anesthesia
  complications of spinal anesthesia will be evaluated, during spinal anesthesia and during the first week

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Kılıç Yılmaz, Study Chair — Trabzon Kanuni Eğitim araştırma Hastanesi
Locations (1):
- TRABZON, Yomra, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
stated that the personal data will not be shared in the participant consent form in the study design.

REFERENCES:
- See also: 'Comparison of Epidrum, Epi-jet, and Loss of Resistance Syringe Techniques for Identifying the Epidural Space in Obstetric Patients' — http://www.ncbi.nlm.nih.gov/pubmed/28891544
- See also: 'Paramedian technique of spinal anesthesia in elderly patients for hip fracture surgery'. — http://www.ncbi.nlm.nih.gov/pubmed/15808095